CLINICAL TRIAL: NCT04512001
Title: A Randomized, Double-Blind, Multiple-Dose, Parallel-Group, Two-Arm Study to Evaluate the Efficacy, Safety and Immunogenicity of MSB11456 Compared to European Union-approved RoActemra® in Patients With Moderately to Severely Active Rheumatoid Arthritis (APTURA I Study)
Brief Title: MSB11456 in Participants With Moderately to Severely Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FKS456-001; 2019-004369-42 (EudraCT Number)
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Results first posted 2022-10-24 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
Keywords: MSB11456; RoActemra®
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MSB11456 (Experimental)
  Interventions: Drug: MSB11456
- RoActemra® (Active Comparator)
  Interventions: Drug: EU-approved RoActemra

INTERVENTIONS:
Drug: MSB11456 — Participants will receive MSB11456 subcutaneously, once a week.
  Arms: MSB11456
Drug: EU-approved RoActemra — Participants will receive EU-approved RoActemra® subcutaneously, once a week.
  Arms: RoActemra®

SUMMARY:
The purpose of the study is to compare the efficacy, safety and immunogenicity of MSB11456 and EU approved RoActemra® in participants with moderately to severely active rheumatoid arthritis.

Participants will be randomized at the beginning of the Core Treatment Period (Baseline to Week 24) to receive either MSB11456 or EU approved RoActemra® once a week (QW). At the beginning of the Extended Treatment Period (Week 24 to Week 52), participants who received RoActemra® will be re-randomized to either continue receiving RoActemra® QW or switch to receive MSB11456 QW.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥18 years of age.
* Diagnosis of rheumatoid arthritis according to the revised 1987 ACR/European League Against Rheumatism (EULAR) Classification 2010 criteria with disease duration of ≥6 months.
* Have moderately to severely active rheumatoid arthritis.
* Must have been treated with methotrexate for at least 12 consecutive weeks immediately prior to randomization and are on a stable dose between 10 and 25 mg/week methotrexate for the last 8 weeks prior to screening.
* Have had previous inadequate clinical response to at least one modifying anti-rheumatic drug.
* Women of childbearing potential (i.e., considered fertile following menarche and until becoming postmenopausal unless permanently sterile) can participate only if they have a negative serum pregnancy test at screening and a negative urine pregnancy test at Day -1 before randomization. Women of childbearing potential must have used and agree to use a highly effective contraception (i.e., methods with a failure rate of less than 1% per year), for 4 weeks before randomization and must agree to continue to practice adequate contraception for 3 months after the last study drug administration.
* Must voluntarily give written informed consent before any study-related activities are performed. Participants must read and fully understand the Informed Consent Form and the requirements of the study. Participants must be willing to comply with all study visits and assessments. Participants must be willing to complete each study procedure. Note: A separate Informed Consent Form (containing important information about COVID 19, clinical research study participation and participant consent) will be provided to and signed by each participant to provide information on the general risks of study participation related to COVID-19 and to document that it is understood by the participant. Another separate Informed Consent Form will be required to be understood and signed by partners of male participating patients who become pregnant during the study or within 10 weeks after the participating patient's last dose of study drug.

Exclusion Criteria:

* American College of Rheumatology functional class IV as defined by the ACR classification of functional status or wheelchair/bedbound.
* Previously received tocilizumab, an investigational or licensed biosimilar of tocilizumab or any interleukin-6 acting drugs.
* Prior use of targeted synthetic disease-modifying anti-rheumatic drugs like janus kinase inhibitors.
* Prior use of more than 2 biologic treatments for rheumatoid arthritis.
* Received a live or attenuated vaccine within 4 weeks prior to randomization.
* Participant is considered by the Investigator, for any reason, to be an unsuitable candidate for the study. Investigator should specifically evaluate the participant's eligibility taking into consideration COVID-19 risk factors and situation.
* Has a serious and/or unstable and/or poorly controlled medical condition such as but not limited to poorly controlled diabetes, unstable ischemic heart disease, uncontrolled hypertension or other cardiovascular, cerebrovascular, cardiovascular, gastrointestinal disease, hepatic, renal, hematological, endocrine, nervous system or pulmonary disease or other relevant medical condition or a history of clinically significant disease or any other condition that, in the opinion of the Investigator, would put the participant at risk by participation in the study.
* Confirmed or, based on the signs and symptoms observed at the time of assessment, suspected active COVID-19 infection at the time of screening and/or randomization.
* Has had any infection as follows:

  1. Herpes zoster or any opportunistic invasive infection within 6 months of screening.
  2. Frequent, chronic or recurrent infections.
  3. A positive test for human immunodeficiency virus subtype 1 (HIV-1) or 2 (HIV-2), hepatitis C antibody, hepatitis B surface antigen and/or core antibody for immunoglobulin G and/or immunoglobulin M or total immunoglobulin at screening.
  4. A serious infection within 8 weeks prior to randomization.
  5. Required treatment with oral antibiotics and/or anti-fungal drugs within 14 days prior to randomization.
* Medical evidence of active or latent tuberculosis as indicated by a positive QuantiFERON®-TB Gold Plus test, chest X-ray and/or clinical examination or has had active or latent tuberculosis disease at any time in the past.
* Received a COVID 19 vaccine within 4 weeks prior to randomization, are receiving ongoing COVID-19 vaccination at the time of screening or plan to receive COVID-19 vaccination before the completion of the Week 30 visit of the study. COVID-19 vaccination is considered ongoing if a multidose regimen has been started but has not been completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (85):
- Bulgaria (10):
  - Medical Center Hipokrat 2000 OOD, Haskovo, Haskovo
  - MHAT "Lyulin" EAD, Sofia, Sofia
  - Military Medical Academy - Sofia, Sofia, Sofia
  - Medical Center N.I.Pirogov EOOD, Sofia, Sofia
  - Medical Center MedConsult Pleven, Pleven
  - University Multiprofile Hospital for Active Treatment Pulmed, Plovdiv
  - Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Medical Center Teodora, Rousse
  - Diagnostic and Consultative Center Equita, Varna
  - MC Sanador M, Vidin
- Czechia (8):
  - Revmatologie, s.r.o., Brno, Jihormoravsky KRAJ
  - Medical Plus, Uherské Hradiště, Jihormoravsky KRAJ
  - Revmatologie MUDr. Zuzana Urbanova, Prague, Prague
  - CCR Ostrava, Ostrava, Severomoravsky KRAJ
  - Revmatologie MUDr. Klára Šírová s.r.o., Ostrava, Severomoravsky KRAJ
  - PV-Medical Services, s.r.o., Zlín, Severomoravsky KRAJ
  - Vesalion s.r.o., Ostrava
  - Revmatologicky Ustav, Prague
- Georgia (9):
  - Helsicore - Israeli Georgian Medical Research Clinic, Tbilisi
  - Research Institute of Clinical Medicine, Tbilisi
  - The First University Clinic, Tbilisi
  - EVEX Hospitals - Caraps Medline, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
  - MediClub Georgia, Tbilisi
  - Georgian Dutch Hospital Ltd, Tbilisi
  - Mtskheta Street Clinic, Tbilisi
  - Tbilisi Heart Center, Tbilisi
- Hungary (8):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes, Csongrád megye
  - DRC Gyogyszervizsgalo Kozpont Kft., Székesfehérvár, Fejér
  - SALDINVEST Befektetesi es Vagyonkezelo Korlatolt Felelossegu Tarsasag, Székesfehérvár, Fejér
  - Integrity Gyogyaszati Kozpont, Zalaegerszeg, Zala County
  - Revita Reumatologiai Rendelo, Budapest
  - MÁV Kórház és Rendelőintézet Rheumatológia, Szolnok
  - Vital Medical Center Orvosi es Fogaszati Kozpont, Veszprém
- Moldova (4):
  - Institutia Medico-Sanitara Publica Institutul de Cardiologie, Chisinau
  - Spitalul Clinic Republican, Chisinau
  - IMSP Spitalul Clinic Municipal Sfanta Treime, Chisinau
  - Instituţia Medico-Sanitară Publică Institutul de Cardiologie, Chisinau
- Poland (27):
  - Solumed Centrum Medyczne, Poznan, Greater Poland Voivodeship
  - Centrum Badan Klinicznych S.C., Poznan, Greater Poland Voivodeship
  - Ai Centrum Medyczne, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne HCP, Poznan, Greater Poland Voivodeship
  - Nasz Lekarz Osrodek Badan Klinicznych - Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Nasz Lekarz Przychodnie Medyczne, Torun, Kuyavian-Pomeranian Voivodeship
  - Grazyna Pulka Specjalistyczny Osrodek All-med, Krakow, Lesser Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - WroMedica, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne Oporow, Wroclaw, Lower Silesian Voivodeship
  - Samodzielny Publiczny Zespol Opieki Zdrowotnej w Tomaszow Lubelski, Tomaszów Lubelski, Lublin Voivodeship
  - Twoja Przychodnia-Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - RCMed Oddzial Sochaczew, Sochaczew, Masovian Voivodeship
  - Medycyna Kliniczna, Warsaw, Masovian Voivodeship
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw, Masovian Voivodeship
  - Ars Rheumatica - Reumatika Centrum Reumatologii, Warsaw, Masovian Voivodeship
  - Barwijuk Clinics, Warsaw, Masovian Voivodeship
  - Centrum Medyczne AMED Warszawa Targowek, Warsaw, Masovian Voivodeship
  - SANUS Szpital Specjalistyczny, Stalowa Wola, Podkarpackie Voivodeship
  - Osteo-Medic, Bialystok, Podlaskie Voivodeship
  - ClinicMed Daniluk Nowak Spolka Jawna, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia w Gdyni, Gdynia, Pomeranian Voivodeship
  - Silmedic w Swidniku, Katowice, Silesian Voivodeship
  - Ambulatorium Sp. z, Elblag, Warmian-Masurian Voivodeship
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag, Warmian-Masurian Voivodeship
  - Centrum Terapii Wspolczesnej, Lodz, Łódź Voivodeship
  - TRIALMED CRS Piotrków Trybunalski, Piotrkow Trybunalski, Łódź Voivodeship
- Russia (12):
  - Clinical Rheumatological Hospital Number 25, Saint Petersburg, Sankt-Peterburg
  - Kazan State Medical University, Kazan', Tatarstan Republic
  - State Budgetary Healthcare Institution of the Yaroslavl Region Clinical Hospital No. 2, Yaroslavl, Yaroslavlr
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - Medical Center Revma-Med, Kemerovo
  - NIARMEDIK - Clinic on Clinic on Kitai Gorod, Moscow
  - Medical Center Health Family, Novosibirsk
  - Polyclinic of Private Security Personnel, Saint Petersburg
  - Saratov Regional Clinical Hospital, Saratov
  - Departmental Hospital at Smolensk Station of JSC RZhD, Smolensk
  - Biomed, Vladimir
  - CjSC "Center of Family Medicine", Yekaterinburg
- Serbia (4):
  - Institute of Rheumatology, Belgrade
  - Institut za Lecenje i Rehabilitaciju Niška Banja, Niška Banja
  - Specijalna Bolnica za Reumatske bolesti Novi Sad, Novi Sad
  - General Hospital Djordje Jovanovic Zrenjanin, Zrenjanin
- Slovakia (3):
  - REUMEX s.r.o., Rimavská Sobota
  - LERAM s.r.o., Topoľčany
  - ALBAMED s.r.o., Zvolen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zubrzycka-Sienkiewicz A, Klama K, Ullmann M, Petit-Frere C, Baker P, Monnet J, Illes A. Comparison of the efficacy and safety of a proposed biosimilar MSB11456 with tocilizumab reference product in subjects with moderate-to-severe rheumatoid arthritis: results of a randomised double-blind study. RMD Open. 2024 Feb 5;10(1):e003596. doi: 10.1136/rmdopen-2023-003596. PMID 38316489

RESULTS

PARTICIPANT FLOW:
Groups:
- Core Treatment Period: MSB11456: Participants received MSB11456 subcutaneously, once a week during the core treatment period (Baseline to Week 24).
- Core Treatment Period: RoActemra®: Participants received EU-approved RoActemra® subcutaneously, once a week during the core treatment period (Baseline to Week 24).
- Core Treatment Period: MSB11456; Extended Treatment Period: MSB11456: Participants who received MSB11456 during the core treatment period (Baseline to Week 24). Participants were then re-randomized to continue receiving MSB11456 subcutaneously, once a week for an additional 28-week during the extended treatment period (Week 24 to Week 52).
- Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456: Participants who received EU-approved RoActemra® during the core treatment period (Baseline to Week 24).
  Participants were then re-randomized to begin receiving MSB11456 subcutaneously, once a week for an additional 28-week during the extended treatment period (Week 24 to Week 52).
- Core Treatment Period: EU-approved RoActemra®; Extended Treatment Period: EU-approved RoActemra®: Participants who received EU-approved RoActemra® during the core treatment period (Baseline to Week 24).
  Participants were then re-randomized to continue receiving EU-approved RoActemra® subcutaneously, once a week for an additional 28-week during the extended treatment period (Week 24 to Week 52).
Period: Week 0 to Week 24
Arm/Group | Core Treatment Period: MSB11456 | Core Treatment Period: RoActemra® | Core Treatment Period: MSB11456; Extended Treatment Period: MSB11456 | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 | Core Treatment Period: EU-approved RoActemra®; Extended Treatment Period: EU-approved RoActemra®
Started | 302 | 302 | 0 | 0 | 0
Received Treatment | 302 | 302 | 0 | 0 | 0
Completed (Re-randomized at Week 24) | 267 | 276 | 0 | 0 | 0
Not Completed | 35 | 26 | 0 | 0 | 0
Not completed — Adverse Event | 14 | 10 | 0 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 9 | 0 | 0 | 0
Not completed — Discontinued treatment prior to Week 24 | 4 | 4 | 0 | 0 | 0
Not completed — Withdrawal By Sponsor's Decision | 1 | 0 | 0 | 0 | 0
Not completed — Subject Did Not Meet Eligibility But Was Randomized | 0 | 1 | 0 | 0 | 0
Period: Week 24 to Week 63
Arm/Group | Core Treatment Period: MSB11456 | Core Treatment Period: RoActemra® | Core Treatment Period: MSB11456; Extended Treatment Period: MSB11456 | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 | Core Treatment Period: EU-approved RoActemra®; Extended Treatment Period: EU-approved RoActemra®
Started | 0 | 0 | 267 | 139 | 137
Received Treatment | 0 | 0 | 266 | 139 | 136
Completed | 0 | 0 | 244 | 123 | 122
Not Completed | 0 | 0 | 23 | 16 | 15
Not completed — Adverse Event | 0 | 0 | 13 | 8 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 4 | 6
Not completed — Miscellaneous | 0 | 0 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) Analysis Set: includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Treatment Period: MSB11456 | Core Treatment Period: RoActemra® | Total
Number analyzed (Participants) | 302 | 302 | 604
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (12.72) | 53.2 (11.33) | 52.2 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 248 | 498
  Male | 52 | 54 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 300 | 300 | 600
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 302 | 302 | 604
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 19 | 23 | 42
  Czechia | 19 | 25 | 44
  Poland | 156 | 147 | 303
  Moldova | 14 | 9 | 23
  Georgia | 43 | 51 | 94
  Slovakia | 5 | 1 | 6
  Bulgaria | 18 | 16 | 34
  Serbia | 7 | 11 | 18
  Russia | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS28-ESR)
Description: The DAS28-ESR is a measure of disease activity in 28 joints that consists of a composite numerical score of the following variables: Tender Joint Count (TJC), Swollen Joint Count (SJC), erythrocyte sedimentation rate (ESR) and Patient's Global Assessment of Disease Activity.
  The DAS28-ESR score was derived using the formula: DAS28-ESR = 0.56*√(TJC28) + 0.28*√(SJC28) + 0.014*GH + 0.70*Ln(ESR), where, TJC28 = 28 joint count for tenderness, SJC28 = 28 joint count for swelling, Ln(ESR) = natural logarithm of ESR, GH = the general health component of the DAS (i.e., Patient's Global Assessment of Disease Activity on a scale of 1 to 100 where 100 is maximal activity).
  Higher values mean a higher disease activity. The level of disease activity can be interpreted as:
  * Remission (score of <2.6).
  * Low (score of ≤2.6 to <3.2).
  * Moderate (score of ≤3.2 to ≤5.1).
  * High (score of >5.1)
  A negative change from baseline indicates an improvement.
Time Frame: Baseline; Week 24
Population: ITT Analysis Set: includes all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Core Treatment Period: MSB11456 | Core Treatment Period: RoActemra®
Number analyzed (Participants) | 302 | 302
score on a scale | -3.53 (0.106) | -3.54 (0.106)
Statistical Analysis 1: Comparison: Core Treatment Period: MSB11456 vs Core Treatment Period: RoActemra®; Test type: Equivalence — Margins for results to be considered equivalent: -0.6 to 0.5; Least squares means difference = 0.01, 90% CI 2-sided [-0.16 to 0.18]

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS28-ESR)
Description: The DAS28-ESR is a measure of disease activity in 28 joints that consists of a composite numerical score of the following variables: TJC, SJC, ESR and Patient's Global Assessment of Disease Activity.
  The DAS28-ESR score was derived using the formula: DAS28-ESR = 0.56*√(TJC28) + 0.28*√(SJC28) + 0.014*GH + 0.70*Ln(ESR), where, TJC28 = 28 joint count for tenderness, SJC28 = 28 joint count for swelling, Ln(ESR) = natural logarithm of ESR, GH = the general health component of the DAS (i.e., Patient's Global Assessment of Disease Activity on a scale of 1 to 100 where 100 is maximal activity).
  Higher values mean a higher disease activity. The level of disease activity can be interpreted as:
  * Remission (score of <2.6).
  * Low (score of ≤2.6 to <3.2).
  * Moderate (score of ≤3.2 to ≤5.1).
  * High (score of >5.1)
  A negative change from baseline indicates an improvement. For weeks 30, 42 and 52, the extended baseline (week 24) was used for the change in DAS28-ESR calculation.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16; Extended Period Baseline (Week 24), Week 30, Week 42, and Week 52
Population: ITT Analysis Set: includes all randomized participants in either the Core Treatment period or the Extended Treatment period and who had a result at baseline and at each specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Core Treatment Period: MSB11456; Extended Treatment Period: MSB11456: Participants received MSB11456 subcutaneously, once a week during the core treatment period (Baseline to Week 24). Participants were then re-randomized to continue receiving MSB11456 subcutaneously, once a week during the extended treatment period (Week 24 to Week 52).
- Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456: Participants received EU-approved RoActemra® subcutaneously, once a week during the core treatment period (Baseline to Week 24). Participants were then re-randomized to begin receiving MSB11456 subcutaneously, once a week during the extended treatment period (Week 24 to Week 52).
- Core Treatment Period: EU-approved RoActemra®; Extended Treatment Period: EU-approved RoActemra®: Participants received EU-approved RoActemra® subcutaneously, once a week during the core treatment period (Baseline to Week 24). Participants were then re-randomized to continue receiving EU-approved RoActemra® subcutaneously, once a week during the extended treatment period (Week 24 to Week 52).
Arm/Group | Core Treatment Period: MSB11456 | Core Treatment Period: RoActemra® | Core Treatment Period: MSB11456; Extended Treatment Period: MSB11456 | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 | Core Treatment Period: EU-approved RoActemra®; Extended Treatment Period: EU-approved RoActemra®
Number analyzed (Participants) | 302 | 302 | 267 | 139 | 137
score on a scale
  Week 2: number analyzed (Participants) | 288 | 295 | 0 | 0 | 0
  Week 2 | -1.24 (1.022) | -1.21 (0.949) |  |  |
  Week 4: number analyzed (Participants) | 294 | 297 | 0 | 0 | 0
  Week 4 | -1.96 (1.184) | -1.98 (1.135) |  |  |
  Week 8: number analyzed (Participants) | 286 | 293 | 0 | 0 | 0
  Week 8 | -2.75 (1.220) | -2.69 (1.260) |  |  |
  Week 12: number analyzed (Participants) | 282 | 292 | 0 | 0 | 0
  Week 12 | -3.13 (1.249) | -3.09 (1.279) |  |  |
  Week 16: number analyzed (Participants) | 282 | 292 | 0 | 0 | 0
  Week 16 | -3.41 (1.288) | -3.32 (1.242) |  |  |
  Week 30: number analyzed (Participants) | 0 | 0 | 261 | 136 | 133
  Week 30 |  |  | -0.16 (0.801) | -0.13 (0.756) | -0.02 (0.863)
  Week 42: number analyzed (Participants) | 0 | 0 | 258 | 134 | 132
  Week 42 |  |  | -0.34 (1.042) | -0.08 (1.026) | -0.27 (1.031)
  Week 52: number analyzed (Participants) | 0 | 0 | 248 | 126 | 126
  Week 52 |  |  | -0.42 (1.185) | -0.31 (1.064) | -0.37 (1.086)

3. Secondary Outcome: Number of Participants With 20% Improvement in American College of Rheumatology (ACR20) Response
Description: ACR20 was defined as the number of participants with at least 20% improvement from baseline in number of tender and swollen joints (68/66 joint count), and at least 20% improvement from baseline in three or more of the 5 ACR Core Set measures:
  * Patient's Assessment of Arthritis Pain
  * Physical Function Assessment (Health Assessment Questionnaire-Disability Index)
  * Acute phase reactant level (erythrocyte sedimentation rate or C-reactive protein)
  * Patient's Global Assessment of Disease Activity and
  * Physician's Global Assessment of Disease Activity
Time Frame: Baseline; Week 24
Population: ITT Analysis Set: includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Core Treatment Period: MSB11456 | Core Treatment Period: RoActemra®
Number analyzed (Participants) | 302 | 302
Participants | 244 | 256
Statistical Analysis 1: Comparison: Core Treatment Period: MSB11456 vs Core Treatment Period: RoActemra®; Test type: Equivalence — Margins for results to be considered equivalent: -15%, 15%; Difference in % Response Rate = -3.94, 95% CI 2-sided [-9.97 to 2.11]

4. Secondary Outcome: Number of Participants Who Experienced One or More Treatment-Emergent Adverse Event (TEAE)
Time Frame: Baseline to end of study, up to Week 63
Population: Safety Analysis Set: all participants who received at least one dose of study drug (MBS11456 or EU-approved RoActemra).
Measure: Count of Participants; unit: Participants
Groups:
- MSB11456: All participants who received MSB11456 at any time in either the Core Treatment Period (Baseline to Week 24) and/or the Extended Treatment Period (Week 24 to Week 52).
  Participants received MSB11456 subcutaneously, once a week.
- EU-approved RoActemra®: All participants who only received EU-approved RoActemra® during the Core Treatment Period (Baseline to Week 24) and/or the Extended Treatment Period (Week 24 to Week 52).
  Participants received EU-approved RoActemra® subcutaneously, once a week.
Arm/Group | MSB11456 | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 | EU-approved RoActemra®
Number analyzed (Participants) | 302 | 139 | 163
Participants | 237 | 105 | 125

5. Secondary Outcome: Number of Participants Who Experienced One or More Treatment-Emergent Serious Adverse Event (TESAE)
Time Frame: Baseline to end of study, up to Week 63
Population: Safety Analysis Set: all participants who received at least one dose of study drug (MBS11456 or EU-approved RoActemra).
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11456 | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 | EU-approved RoActemra®
Number analyzed (Participants) | 302 | 139 | 163
Participants | 51 | 20 | 33

6. Secondary Outcome: Percentage of Participants With Positive Anti-Drug Antibodies (ADAs)
Time Frame: Baseline, Week 2, Week 12, Week 24, Week 30, Week 52 and Week 55
Population: All participants who received at least one dose of study drug (MBS11456 or EU-approved RoActemra) in either the Core Treatment Period or the Extended Treatment Period and had a valid ADA result at the specific time points.
Measure: Number; unit: percentage of participants
Arm/Group | Core Treatment Period: MSB11456 | Core Treatment Period: RoActemra® | Core Treatment Period: MSB11456; Extended Treatment Period: MSB11456 | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 | Core Treatment Period: EU-approved RoActemra®; Extended Treatment Period: EU-approved RoActemra®
Number analyzed (Participants) | 302 | 302 | 266 | 139 | 136
percentage of participants
  Overall (includes all time points expect Baseline): number analyzed (Participants) | 299 | 301 | 265 | 137 | 135
  Overall (includes all time points expect Baseline) | 96.0 | 96.3 | 97.4 | 97.1 | 94.1
  Baseline: number analyzed (Participants) | 302 | 302 | 0 | 0 | 0
  Baseline | 6.6 | 8.3 |  |  |
  Week 2: number analyzed (Participants) | 287 | 291 | 0 | 0 | 0
  Week 2 | 87.1 | 88.7 |  |  |
  Week 12: number analyzed (Participants) | 281 | 292 | 0 | 0 | 0
  Week 12 | 79.0 | 74.3 |  |  |
  Week 24 (Extended Treatment Period Baseline): number analyzed (Participants) | 274 | 283 | 266 | 139 | 136
  Week 24 (Extended Treatment Period Baseline) | 76.3 | 68.6 | 86.8 | 77.7 | 87.5
  Week 30: number analyzed (Participants) | 0 | 0 | 262 | 134 | 132
  Week 30 |  |  | 76.7 | 73.1 | 65.9
  Week 52: number analyzed (Participants) | 0 | 0 | 246 | 125 | 126
  Week 52 |  |  | 80.9 | 76.8 | 61.1
  Week 55: number analyzed (Participants) | 0 | 0 | 242 | 122 | 122
  Week 55 |  |  | 81.4 | 82.8 | 77.9

7. Secondary Outcome: Anti-Drug Antibodies (ADAs) Titer Levels
Time Frame: Baseline, Week 2, Week 12, Week 24, Week 30, Week 52 and Week 55
Population: as for outcome 6
Measure: Geometric Mean (Full Range); unit: titer
Arm/Group | Core Treatment Period: MSB11456 | Core Treatment Period: RoActemra® | Core Treatment Period: MSB11456; Extended Treatment Period: MSB11456 | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 | Core Treatment Period: EU-approved RoActemra®; Extended Treatment Period: EU-approved RoActemra®
Number analyzed (Participants) | 302 | 302 | 266 | 139 | 136
titer
  Overall (includes all time points except Baseline): number analyzed (Participants) | 299 | 301 | 265 | 137 | 135
  Overall (includes all time points except Baseline) | 106.3 [60 to 15360] | 104.0 [60 to 122880] | 215.4 [60 to 15360] | 166.3 [60 to 15360] | 101.1 [60 to 960]
  Baseline: number analyzed (Participants) | 302 | 302 | 0 | 0 | 0
  Baseline | 71.4 [60 to 960] | 130.4 [60 to 1920] |  |  |
  Week 2: number analyzed (Participants) | 287 | 291 | 0 | 0 | 0
  Week 2 | 81.2 [60 to 1920] | 88.1 [60 to 15360] |  |  |
  Week 12: number analyzed (Participants) | 281 | 292 | 0 | 0 | 0
  Week 12 | 113.8 [60 to 960] | 123.1 [60 to 122880] |  |  |
  Week 24 (Extended Treatment Period Baseline): number analyzed (Participants) | 274 | 283 | 266 | 139 | 136
  Week 24 (Extended Treatment Period Baseline) | 138.4 [60 to 15360] | 102.9 [60 to 1920] | 127.7 [60 to 15360] | 106.1 [60 to 1920] | 95.6 [60 to 960]
  Week 30: number analyzed (Participants) | 0 | 0 | 262 | 134 | 132
  Week 30 |  |  | 173.0 [60 to 15360] | 130.6 [60 to 7680] | 93.7 [60 to 960]
  Week 52: number analyzed (Participants) | 0 | 0 | 246 | 125 | 126
  Week 52 |  |  | 230.9 [60 to 7680] | 174.7 [60 to 15360] | 96.7 [60 to 480]
  Week 55: number analyzed (Participants) | 0 | 0 | 242 | 122 | 122
  Week 55 |  |  | 251.2 [60 to 15360] | 200.8 [60 to 15360] | 112.4 [60 to 480]

8. Secondary Outcome: Percentage of Participants With Neutralizing Antibodies (NAb)
Time Frame: Baseline, Week 2, Week 12, Week 24, Week 30, Week 52 and Week 55
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Core Treatment Period: MSB11456 | Core Treatment Period: RoActemra® | Core Treatment Period: MSB11456; Extended Treatment Period: MSB11456 | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 | Core Treatment Period: EU-approved RoActemra®; Extended Treatment Period: EU-approved RoActemra®
Number analyzed (Participants) | 302 | 302 | 266 | 139 | 136
percentage of participants
  Overall (includes all time points except Baseline): number analyzed (Participants) | 299 | 301 | 265 | 137 | 135
  Overall (includes all time points except Baseline) | 8.4 | 11.3 | 13.2 | 16.8 | 11.9
  Baseline: number analyzed (Participants) | 302 | 302 | 0 | 0 | 0
  Baseline | 0 | 0 |  |  |
  Week 2: number analyzed (Participants) | 287 | 291 | 0 | 0 | 0
  Week 2 | 3.8 | 3.4 |  |  |
  Week 12: number analyzed (Participants) | 281 | 292 | 0 | 0 | 0
  Week 12 | 2.5 | 4.1 |  |  |
  Week 24 (Extended Treatment Period Baseline): number analyzed (Participants) | 274 | 283 | 266 | 139 | 136
  Week 24 (Extended Treatment Period Baseline) | 2.9 | 4.9 | 3.8 | 5.8 | 5.9
  Week 30: number analyzed (Participants) | 0 | 0 | 262 | 134 | 132
  Week 30 |  |  | 6.1 | 9.7 | 3.0
  Week 52: number analyzed (Participants) | 0 | 0 | 246 | 125 | 126
  Week 52 |  |  | 1.6 | 2.4 | 1.6
  Week 55: number analyzed (Participants) | 0 | 0 | 242 | 122 | 122
  Week 55 |  |  | 7.0 | 6.6 | 9.0

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 63
Description: Safety Analysis Set: all participants who received at least one dose of study drug (MBS11456 or EU-approved RoActemra). The tables below only include treatment-emergent adverse events and "Other Adverse Events" only include non-serious TEAEs.
Groups:
- MSB11456: All participants who received MSB11456 in the Core Treatment Period (Baseline to Week 24) and who could then be re-randomized to continue MSB11456 in the Extended Treatment Period (Week 24 to Week 52).
- EU-approved RoActemra®: All participants who received EU-approved RoActemra® in the Core Treatment Period (Baseline to Week 24) and who could then re-randomized to continue RoActemra® in the Extended Treatment Period (Week 24 to Week 52).
Arm/Group | MSB11456 | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 | EU-approved RoActemra®
All-Cause Mortality (participants affected / at risk) | 0/302 | 1/139 | 3/163
Serious Adverse Events (participants affected / at risk) | 51/302 | 20/139 | 33/163
Other Adverse Events (participants affected / at risk) | 163/302 | 82/139 | 92/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSB11456 (N=302) | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 (N=139) | EU-approved RoActemra® (N=163)
COVID-19 (Infections and infestations) | 38 | 12 | 19
Abscess limb (Infections and infestations) | 1 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery disease (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MSB11456 (N=302) | Core Treatment Period: RoActemra®; Extended Treatment Period: MSB11456 (N=139) | EU-approved RoActemra® (N=163)
Alanine aminotransferase increased (Investigations) | 36 | 22 | 22
Aspartate aminotransferase increased (Investigations) | 19 | 9 | 10
Leukopenia (Blood and lymphatic system disorders) | 22 | 8 | 12
Neutropenia (Blood and lymphatic system disorders) | 19 | 8 | 10
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 5 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 2 | 7
Blood bilirubin increased (Investigations) | 11 | 8 | 3
Mycobacterium tuberculosis complex test positive (Investigations) | 14 | 4 | 4
Blood pressure increased (Investigations) | 6 | 4 | 6
Blood bilirubin unconjugated increased (Investigations) | 5 | 5 | 4
Blood cholesterol increased (Investigations) | 4 | 4 | 3
Gamma-glutamyltransferase increased (Investigations) | 5 | 2 | 4
Low density lipoprotein increased (Investigations) | 5 | 4 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 4
COVID-19 (Infections and infestations) | 38 | 12 | 19
Upper respiratory tract infection (Infections and infestations) | 17 | 6 | 10
Nasopharyngitis (Infections and infestations) | 9 | 5 | 9
Urinary tract infection (Infections and infestations) | 5 | 4 | 3
Bronchitis (Infections and infestations) | 7 | 0 | 3
Pharyngitis (Infections and infestations) | 2 | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 5 | 6 | 2
Lymphopenia (Blood and lymphatic system disorders) | 5 | 1 | 4
Nausea (Gastrointestinal disorders) | 9 | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 | 5 | 5
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 | 4 | 4
Headache (Nervous system disorders) | 17 | 2 | 4
Dizziness (Nervous system disorders) | 4 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Hypertension (Vascular disorders) | 13 | 6 | 4
Cystitis noninfective (Renal and urinary disorders) | 2 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT04512001/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT04512001/SAP_001.pdf